CLINICAL TRIAL: NCT04522635
Title: Fluid Mobilization in Hospitalized Patients With Acute Kidney Injury
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Grifols Biologicals, LLC (Industry)
Responsible Party: Principal Investigator, Ravindra Mehta, Professor Emeritus, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 141779
Record Dates: First submitted 2020-08-18; First posted 2020-08-21 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Hypotension During Dialysis; Fluid Overload
MeSH Terms: conditions — Edema | interventions — Albumins

STUDY DESIGN:
Intervention Model Description: Patients will be randomized for a minimum of 4 and maximum of 6 consecutive dialysis sessions to one of two sequences:
  1. Sequence A: Albumin in sessions 1, 3 and 5 and saline in sessions 2, 4 and 6
  2. Sequence B: Saline in sessions 1, 3, 5 and albumin in sessions 2, 4 and 6 Dialysis Procedures (Standard of Care with the exception of Albumin which is additional and for research purposes only): All dialysis sessions will include standard procedures and monitoring. Dialysis prescriptions will be individualized for each patient and will be maintained through each of the 6 sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- albumin (Active Comparator): albumin (100 ml of Grifols 25%) given intravenously at the start of IHD
  Interventions: Drug: (100 ml of Albumin 25%)
- normal saline (Placebo Comparator): 0.9% sodium chloride (normal saline (NS)) given intravenously at the start of IHD
  Interventions: Drug: (100 ml of Albumin 25%)

INTERVENTIONS:
Drug: (100 ml of Albumin 25%) — single dose of 25g albumin (100 ml of Grifols 25%) given intravenously at the start of IHD
  Other Names: albumin

SUMMARY:
Hospitalized patients often suffer from an acute shutdown of kidney function secondary to infections, use of antibiotics, or use of intravenous contrast agents. This results in the accumulation of toxic substances and retention of fluid in the body. Dialysis techniques are often needed to manage these patients to remove the retained toxic substances and extra fluid and allow the kidney time to recover. The amount and duration of fluid accumulation have been associated with a higher risk of death and longer hospital stays. Correction of fluid overload with dialysis has been shown to be beneficial in improving the outcomes from these patients. Most patients are quite sick and often have low levels of a blood protein called albumin that makes them more prone to developing low blood pressure during dialysis and limits the ability of dialysis to remove solutes and fluid adequately. Often dialysis sessions are complicated by the development of low blood pressures and symptoms such as nausea, vomiting, and headaches that further compromises dialysis efficacy. In this study, the hypothesis that addition of intravenous albumin during the dialysis session will improve the ability to remove fluid and reduce the incidence of low blood pressure during dialysis thereby improving patient tolerance and the efficacy of the procedure will be tested. Patients with acute kidney failure or end-stage Renal Disease who need dialysis for fluid removal will be allocated to receive albumin or saline as intravenous fluids during individual dialysis sessions and information on how much fluid can be removed and how many complications occur in each session will be recorded. Dialysis sessions with albumin will be compared with those with saline alone to determine the benefit of adding albumin to the treatment. Information obtained from this study will allow physicians to manage patients requiring dialysis for acute kidney failure more effectively and help improve outcomes.

DETAILED DESCRIPTION:
This study will address the following questions:

AIM 1: Can the utilization of intravenous albumin enhance the efficacy of fluid removal in hospitalized patients undergoing dialysis for AKI or ESRD.

The hypothesis to be tested:

1. Addition of albumin solutions to dialysis therapy will enhance the efficacy of fluid removal (total amount of fluid removed)
2. Albumin solutions will improve the efficiency of fluid removal by dialysis per unit time
3. Albumin addition will reduce the time to achieving and maintaining fluid balance and correcting fluid overload.

AIM 2: Can the utilization of IV albumin improve the safety of fluid removal during dialysis?

The hypothesis to be tested:

1. Addition of albumin solutions will reduce the frequency of Intradialytic hypotension associated with fluid removal on dialysis.
2. Albumin solutions given during dialysis will reduce the incidence and magnitude of myocardial stunning associated with fluid removal on dialysis
3. Albumin solutions given during dialysis will reduce post-dialysis symptoms AIM 3: Does utilization of IV albumin improve the microcirculation in hospitalized patients undergoing fluid removal with dialysis?

The hypothesis to be tested:

1. Patients with AKI or ESRD will have deranged microcirculatory profile as compared to normal
2. During fluid removal with dialysis changes in microcirculation correlate with alterations in hemodynamics related to the rate and amount of fluid removal
3. Utilization of IV albumin during dialysis will reduce the microcirculatory stress of fluid removal

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years old
* need for intermittent hemodialysis during hospitalization
* hypoalbuminemia (albumin<3g/dl)

Exclusion Criteria:

* allergy to the components of albumin

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2015-06-03 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
fluid removal | during procedure
  achieved fluid removal expressed as ml/kg/hour

SECONDARY OUTCOMES:
hypotension | during procedure
  cardiovascular complications, including hypotensive episodes

CONTACTS AND LOCATIONS:
Overall Officials: Ravindra L Mehta, MD, Principal Investigator — UCSD

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Macedo E, Karl B, Lee E, Mehta RL. A randomized trial of albumin infusion to prevent intradialytic hypotension in hospitalized hypoalbuminemic patients. Crit Care. 2021 Jan 6;25(1):18. doi: 10.1186/s13054-020-03441-0. PMID 33407747